CLINICAL TRIAL: NCT03028233
Title: Healthy Kids & Families: Overcoming Social, Environmental and Family Barriers to Childhood Obesity Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Oak Hill Community Development Corporation (Unknown); Worcester Public Schools (Unknown)
Responsible Party: Principal Investigator, Milagros Rosal, Professor, University of Massachusetts, Worcester
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H00005048; U48DP005031 (NIH)
Record Dates: First submitted 2017-01-10; First posted 2017-01-23 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Obesity
Keywords: physical activity; healthy eating; weight; families; Community Health Worker; childhood obesity; built environment
MeSH Terms: conditions — Obesity; Motor Activity; Body Weight; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Lifestyles (Experimental): The study will test the impact of a community health worker (CHW)-delivered intervention aimed at helping families overcome barriers to childhood obesity prevention. Barriers include social, environmental, and family issues.
  Interventions: Behavioral: Healthy Lifestyle
- Positive Parenting (Active Comparator): The control condition consists of a community health worker (CHW)-delivered intervention aimed at helping families improve positive parenting skills.
  Interventions: Behavioral: Positive Parenting

INTERVENTIONS:
Behavioral: Healthy Lifestyle — A Community Health Worker coaches families regarding healthy eating, physical activity, and obesity prevention, and promotes the use of existing built environment resources.
  Arms: Healthy Lifestyles
Behavioral: Positive Parenting — A Community Health Worker coaches parents on improving positive parenting skills and promotes the use of relevant community resources.
  Arms: Positive Parenting

SUMMARY:
The study will test the impact of a community health worker (CHW)-delivered intervention aimed at helping families overcome barriers to childhood obesity prevention. Barriers include social, environmental, and family issues.

This intervention will be compared to a control condition consisting of a community health worker (CHW)-delivered intervention aimed at helping families improve positive parenting skills.

DETAILED DESCRIPTION:
The study will test the impact of a community health worker (CHW)-delivered intervention aimed at helping families overcome barriers to childhood obesity prevention. Barriers include social, environmental, and family issues.

This intervention will be compared to a control condition consisting of a community health worker (CHW)-delivered intervention aimed at helping families improve positive parenting skills.

The intervention uses multiple delivery modalities to maintain novelty and prevent attrition/burden. These include home visits, telephone contacts, print (literacy sensitive newsletters), social media (Facebook), and community events. Parents and children will complete scheduled assessments at baseline, 6-, 12-, 18- and 24-month follow-up.

The Specific Aims are:

Aim 1: To determine the effectiveness of the intervention compared to the control condition on child physical activity, healthy eating, BMI and utilization of built environment resources.

Aim 2: To determine the effectiveness of the intervention compared to the control condition on parent physical activity, healthy eating, BMI.

Aim 3: To examine the potential scalability of the intervention guided by the RE-AIM (Reach Effectiveness Adoption Implementation Maintenance) model.

ELIGIBILITY:
Inclusion Criteria:

* Eligible individuals for the research study are parents/guardians and their K-6th grade children attending one of 9 schools in the greater Worcester area. Parents and their children are recruited as parent-child dyads.

Exclusion Criteria:

* Has an inability or unwillingness to give informed consent or assent
* Is a prisoner

Exclusion (child only)

* The child has been told by a doctor that they cannot walk or eat fruits and vegetables.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2014-09; Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
child BMI z-score | 2 years
  Weight and height is measured using standard methodology, with children wearing light clothing and no shoes. Weight is measured to the nearest 0.5 lb on a digital scale. Height is measured to the nearest tenth of a centimeter using a stadiometer. BMI is calculated: weight (kg)/height squared (meters) for age and gender using United States Centers for Disease Control and Prevention BMI charts growth charts.

SECONDARY OUTCOMES:
Child Dietary Behaviors: Overall | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration: Selected items from the Massachusetts Parent Child Longitudinal Cohort Survey (Taveras et al., MA-CORD Study Group)
Child Dietary Behaviors for snacks | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration:Snack items from the Beverage and Snack Questionnaire2 (BSQ2) (https://sharedresources.fredhutch.org/documents/beverage-and-snack-questionnaire-2)
Child Dietary Behaviors for Beverages | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration: Beverage Intake Questionnaire (Hedrick et al)
Parent Dietary Behaviors: Overall | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration: Selected items from the Massachusetts Parent Child Longitudinal Cohort Survey (Taveras et al., MA-CORD Study Group)
Parent Dietary Behaviors for Snacks | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration: Snack items from the Beverage and Snack Questionnaire2 (BSQ2) (https://sharedresources.fredhutch.org/documents/beverage-and-snack-questionnaire-2)
Parent Dietary Behaviors for Beverages | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration: Beverage Intake Questionnaire (Hedrick et al)
Child Physical Activity and Sedentariness: Massachusetts Parent Child Longitudinal Cohort Survey | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration: Selected items from the Massachusetts Parent Child Longitudinal Cohort Survey (Taveras et al., MA-CORD Study Group)
Child Physical Activity and Sedentariness: C-PAQ and PAQ-C | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration:Selected items from the Physical Activity C-PAQ (Kemper et al) plus PAQ-C (Kowalski et al) activity questions
Child Physical Activity and Sedentariness: ActiGraph GT1M | 2 years
  Child physical activity and sedentariness are measured by the child wearing the ActiGraph Model GT1M for 7 days averaged. This measure provides data on intensity and duration of activities.
Parent physical activity and sedentariness: Massachusetts Parent Child Longitudinal Cohort Survey | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration:Selected items from the Massachusetts Parent Child Longitudinal Cohort Survey (Taveras et al., MA-CORD Study Group)
Parent physical activity and sedentariness: C-PAQ and PAQ-C | 2 years
  This Outcome Measure is assessed through the following measure, modified for verbal administration: Selected items from the Physical Activity C-PAQ (Kemper et al) plus PAQ-C (Kowalski et al) activity questions
Parent physical activity and sedentariness: ActiGraph GT1M | 2 years
  Parent physical activity and sedentariness are measured by the parent wearing the ActiGraph Model GT1M for 7 days averaged. This measure provides data on intensity and duration of activities
Parent BMI | 2 years
  BMI is calculated with weight and height measurements using standard methodology. Weight is measured to the nearest 0.5 lb on a digital scale. Height is measured to the nearest centimeter using a stadiometer. BMI is calculated: weight (kg)/height squared (meters) for gender using United States Centers for Disease Control and Prevention BMI charts.
Child utilization of built environment resources | 2 years
  Child utilization of built environment resources is assessed by the children wearing a portable GPS unit (~size of a matchbox) when wearing an accelerometer. The GPS unit records the geographic coordinates of the child's activities. Measures of frequency and duration of activities by neighborhood space (e.g., parks) can be ascertained.

CONTACTS AND LOCATIONS:
Overall Officials: Milagros C Rosal, PhD, Principal Investigator — UMass Medical School; Wenjun Li, PhD, Principal Investigator — UMass Medical School
Locations (1):
- UMass Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borg A, Haughton CF, Sawyer M, Lemon SC, Kane K, Pbert L, Li W, Rosal MC. Design and methods of the Healthy Kids & Families study: a parent-focused community health worker-delivered childhood obesity prevention intervention. BMC Obes. 2019 Jun 3;6:19. doi: 10.1186/s40608-019-0240-x. eCollection 2019. PMID 31171975